CLINICAL TRIAL: NCT06421519
Title: Crossover Study of the Work of Breathing at Different Levels of BiPAP Settings in Neonates
Brief Title: Different Levels of BiPAP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRAS 327794
Record Dates: First submitted 2024-05-09; First posted 2024-05-20 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Biphasic continuous positive airway pressure (BiPAP)
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: Infants receive receive three upper pressures of BiPAP: 7, 10 or 13cmH2O for a period of 20 minutes each. Additionally, there will be a control period of 20 minutes between each upper pressure with a baseline pressure constant of 5cmH2O. The order in which they receive the levels of respiratory support will be randomised using an excel random number generator. This allows each infant to be used as their own control, minimising the impact of any underlying confounding factors. The results on each pressure setting will be meaned and compared to each other
Who Masked: Participant, Outcomes Assessor
Masking Description: During the study the infant and their parents will not be aware of which pressures they are on. Due to the nature of the study it is not possible to blind the care provider who in this case is the investigator since they need to manipulate the ventilator settings. However, data analysis with be done using anonymous data and the investigator will be blinded to which pressure settings were used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-term infants requiring primary respiratory support before intubation (Experimental): Infants <34 weeks gestational age who require non-invasive respiratory support who may go on to require invasive ventilation.
  Interventions: Other: BiPAP setting
- Pre-term infants requiring respiratory support after extubation (Experimental): Infants <34 weeks gestational age who were previously invasively ventilated and are currently being weaned onto non-invasive respiratory support and eventually into self-ventilating in room air.
  Interventions: Other: BiPAP setting
- Pre-term infants requiring respiratory support after seven days (Experimental): Infants <34 weeks gestational age who have an ongoing need for non-invasive respiratory support after seven days of life and are likely to develop bronchopulmonary dysplasia.
  Interventions: Other: BiPAP setting

INTERVENTIONS:
Other: BiPAP setting — Infants in this arm of the study will each rotate through three different BiPAP settings. The following BiPAP settings will be used:
  13cmH2O / 5cmH2O, 10cmH2O / 5cmH2O, 7cmH2O / 5cmH2O

SUMMARY:
Some infants with breathing problems at birth may need to be connected to a machine to help support their breathing. The purpose of this study is to optimise the level of breathing support on Bi level continuous airway pressure (BiPAP), a support which gives two levels of support (pressure) to premature infants.

The study is investigating which upper pressure gives the best support, that is results in the baby having to breathe less hard (work of breathing).

Researchers will measure the work of breathing using a small catheter. Infants will receive three different upper pressures of BiPAP with the same baseline pressure for 20 minutes each. In between each upper level they will receive the standard upper pressure for 20 minutes.

DETAILED DESCRIPTION:
Bilevel continuous positive airway pressure (BiPAP) is a type of non-invasive respiratory support which can be used as breathing support in neonates requiring some pressure support to help their breathing. BiPAP provides cycles of higher and lower pressure levels at set intervals, usually with a baseline pressure constant of 5cm H2O.

In the UK, other forms of non-invasive ventilation, such as NIPPV and NIV-NAVA, have been shown to be efficacious, however they are expensive. BiPAP may therefore provide a viable and cost-effective alternative. Currently there are no written guidelines about BiPAP use.

The investigators aim to identify the most efficacious BiPAP settings for preterm infants as primary support and post-extubation as well as in those with evolving BPD. Infants will be studied at three different upper pressure settings for a period of 20 minutes each. The work of breathing will be measured from small pressure transducers situated on a thin catheter, the size of a feeding tube. The catheter will be passed through the mouth and positioned so the tip is in the stomach. Simultaneous measurements for work of breathing using transcutaneous diaphragm electromyography will also be taken. Following the study the infant will subsequently be nursed on the breathing support type associated with the lower work of breathing.

The investigators aim to recruit 21 patients, with 7 in each arm of the trial. Sample size was derived using previous study results in which the SD of the PTPdi was 78cmH2Os/min in 40 preterm infants of 28-34 weeks gestation and a clinically significant difference of 133cmH2Os/min was observed between infants on SNIPPV against high flow NIV support. To detect such a difference with 90% power and 5% significance, 7 infants would be required in each group, that is 21 infants in total in 3 groups.

The parents of potential participants will be approached by the clinical team initially, subsequently the research fellow will provide them with the study information. Responsibility for recording and dating oral, electronic, and written informed consent or advice will be with the researchers identified in the formal delegation log.

Full analyses will be detailed in a statistical analysis plan (SAP), which will be finalised prior to the end of data collection Any exploratory analyses of sub-groups that are of clinical interest will be pre-specified in the SAP. Any deviations from the original SAP will be described and justified in protocol and/or in final report, as appropriate. This trial will be reported according to the CONSORT guidelines for clinical trials (Consolidated Standards Of Reporting Trials statement). Statistical significance will be at 5% level, and analyses will be conducted in STATA. A summary of the planned statistical analysis is included here:

* Descriptive statistics will be used to describe infant demographics. Standard statistical summaries e.g. medians and ranges or means and variances, or proportions and percentages, dependent on the distribution of the outcomes.
* The main analysis will investigate work of breathing at baseline and at each of the 3 upper BiPAP pressure settings. Data will be assessed for normality. If data is not normally distributed, non-parametric statistics will be used. 95% confidence intervals will be reported throughout. Missing data will be described with reasons given where available.

Data collected during the study will be handled and stored in accordance with the General Data Protection Regulation and Data Protection Act (2018), which requires data to be de-identified as soon as it is practical to do so. All data will be completely anonymised for purposes of analysis and any subsequent reports or publications. For the purposes of ongoing data management, once randomised, individual patients will only be identified by trial numbers.

Data will be downloaded from ventilators and pressure transducers to excel using secure password encrypted USB device Data will be uploaded on password protected servers only and anonymised at the point of entry.

Data will be anonymised and identified by a unique identification number (Trial number) only. A trial enrolment log at the sites will list the ID numbers.

Paper study documents will be held at the trial site in a secure location for the duration of the trial. All essential documents will be retained until children reach 25 years old, as per protocol.

A statement of permission to access source data by study staff and for regulatory and audit purposes will be included within the primary care givers consent form with explicit explanation as part of the consent process and Participant Information Sheet.

In principle, anonymised data will be made available for meta-analysis and if requested by other authorised researchers and journals for publication purposes. Requests for access to data will be reviewed by the Chief Investigator.

Each adverse event will be assessed for severity, causality, seriousness and expectedness. All adverse events will be recorded in the medical records in the first instance. All adverse events will be recorded with clinical symptoms and accompanied with a simple, brief description of the event, including dates as appropriate. All serious adverse events will be recorded in the medical records and the CRF.

The Chief Investigator will ensure there are adequate quality and number of monitoring activities conducted by the study team. This will include adherence to the protocol, procedures for consenting and ensure adequate data quality.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born <34 weeks of gestation at KCH requiring primary respiratory support before intubation, after extubation or requiring respiratory support after seven days
* Infants aged between 2 days and 2 months at time of study

Exclusion Criteria:

* Infants with congenital abnormalities of the respiratory system.
* Infants with blood-culture confirmed sepsis.
* Recent gastrointestinal surgery (within 7 days)
* Non-English speakers

Ages: 2 Days to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Work of breathing | Over the last 5 minutes of the 20 minute study period on each setting of BiPAP
  Oesophageal (Poes) and gastric pressures(Pgas) will be measured using a catheter with dual pressure tipped transducers (Gaeltec, Dunvegan, Scotland, UK). Transdiaphragmatic pressure (PTPdi) will be calculated by digital subtraction of the oesophageal from the gastric pressure and tidal volume obtained by digital integration of the flow signal by the acquisition software. The mean PTPdi will be calculated from 20 consecutive breaths to measure work of breathing.
Work of breathing | Over the last 5 minutes of the 20 minute study period on each setting of BiPAP
  Transcutaneous diaphragm electromyography (EMG) will be monitored using a portable 16-channel digital physiological amplifier (Dipha-16; Inbiolab, Groningen, the Netherlands) and three surface electrodes (Kendall H59P cloth electrodes; Covidien, Massachusetts) placed on the infant's abdomen. The device wirelessly transmits to a bedside computer running Polybench (Applied Biosignals, Weener, Germany). Work of breathing will be calculated using the voltages measured from a 5 minute period of recording.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Dassios, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
In principle, anonymised data will be made available for meta-analysis and if requested by other authorised researchers and journals for publication purposes. Requests for access to data will be reviewed by the Chief Investigator.